CLINICAL TRIAL: NCT00893230
Title: A Double-Blind, Randomized, Placebo-Controlled Intervention Study of the Efficacy and Safety of "NFM proBio65" in the Atopic and Allergic Volunteers
Brief Title: A Study of a Probiotic in Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chungbuk National University (Other)
Collaborators: Yeungnam University Hospital (Other); Korea Research Institute of Bioscience & Biotechnology (Other Government); Gachon University Gil Medical Center (Other)
Responsible Party: Youn-Soo Hahn, Department of Pediatrics, College of Medicine, Chungbuk National University, Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS 7403-179
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; chemokines; probiotics
MeSH Terms: conditions — Dermatitis, Atopic | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus sakei KCTC 10755BP (Experimental)
  Interventions: Dietary Supplement: probiotic L sakei KCTC 10755BP
- microcrystalline cellulose (Placebo Comparator)
  Interventions: Dietary Supplement: microcrystalline cellulose (placebo)

INTERVENTIONS:
Dietary Supplement: probiotic L sakei KCTC 10755BP — freeze-dried, 50,0000,0000 colony-forming units, twice daily, for 12 weeks
  Arms: Lactobacillus sakei KCTC 10755BP
Dietary Supplement: microcrystalline cellulose (placebo) — freeze-dried, 50,0000,0000 colony-forming units, twice daily, for 12 weeks
  Arms: microcrystalline cellulose

SUMMARY:
The aim of this study was to assess the clinical effect of Lactobacillus sakei supplementation in children with atopic dermatitis.

DETAILED DESCRIPTION:
Probiotics were also shown to reduce severity of AEDS when administered to infants with early onset AEDS. In contrast, only a few studies have evaluated the therapeutic effectiveness of probiotics on the groups of older children with established AEDS. In these studies, administration of Lactobacillus strains to unselected children aged 1 year and over was associated with improvement in the clinical severity of eczema. The purpose of this study was to evaluate the clinical efficacy in AEDS of a newly identified probiotic strain, Lactobacillus sakei KCTC 10755BP, which showed the most potent inhibitory activity against S aureus growth among Lactobacillus species in our preliminary experiment. We administered L sakei to an unselected group of children aged 2 to 10 years with moderate and severe AEDS and evaluated the clinical outcome at the end of the intervention. In addition, we also measured levels of serum chemokines as activity markers for AEDS to provide a more objective evidence for the beneficial role of this probiotic.

ELIGIBILITY:
Inclusion Criteria:

* patients with atopic dermatitis present for at least 6 months before inclusion
* a total SCORAD score above 25
* a change in a total SCORAD score of not more than 10% within 2 weeks

Exclusion Criteria:

* patients who had been treated with cyclosporine, systemic steroid, topical calcineurin inhibitor, or Chinese herbal medicine during the preceding 3 months

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
SCORAD score | 12 weeks

SECONDARY OUTCOMES:
Chemokine levels | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Youn-Soo Hahn, MD, PhD, Principal Investigator — Department of Pediatrics, College of Medicine and Medical Research Institute, Chungbuk National University, Cheongju, Korea,
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea